CLINICAL TRIAL: NCT00815191
Title: A Comparison Study of the Vital HEAT (vH2) Temperature Management System to Upper-body Forced-air Warming in Patients Undergoing Open Abdominal Surgery Under General Anesthesia
Brief Title: Comparison of Vital HEAT (vH2) Temperature Management System to Upper-body Forced-air Warming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, d sessler, Chairman of Outcomes Research, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 07-1042
Record Dates: First submitted 2008-12-24; First posted 2008-12-29 (Estimated); Results first posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-06

CONDITIONS: Surgery
Keywords: temperature; surgery; heating device

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vital Heat (Active Comparator): Vital HEAT (vH2) Temperature Management System
  Interventions: Device: vital HEAT (vH2) Temperature Management System
- Forced air (Active Comparator): Forced-air warming
  Interventions: Device: a forced-air warming cover

INTERVENTIONS:
Device: a forced-air warming cover — A forced-air warming cover will be placed on the subject prior to surgery, remain on the subject during surgery and removed after surgery.
  Arms: Forced air
Device: vital HEAT (vH2) Temperature Management System — The vital HEAT (vH2) Temperature Management System will be placed on the subjects arm prior to surgery. remain on the arm during surgery and removed after surgery.
  Arms: Vital Heat

SUMMARY:
The primary objective of this study is to determine if the intraoperative distal esophageal (core) temperature with vitalHEAT warming is non-inferior to upper-body forced-air warming in patients undergoing open colectomy under general anesthesia. This is a randomized study.

DETAILED DESCRIPTION:
Participants will be randomized into one of two groups. Patients assigned to vitalHEAT warming will have the circulating-water sleeve applied to an arm that will not require intravenous access. An esophageal temperature probe will be inserted and connected to the anesthesia machine monitoring system. Intravenous fluids will be warmed to 40-42°C.

As soon as practical after induction, the vitalHEAT warmer will be activated in the appropriate patients and set to "high" which is 42°C

An upper-body forced-air warmer will be positioned over the upper body and exposed arms on patients assigned to forced-air heating. The forced air blower will be set to "high" which is 43°C and activated as soon as practical, usually after prepping and draping.

Patients in both groups will be otherwise draped per surgical routine. Ambient temperature will be maintained near 20°C. Active warming will be maintained until just before extubation. The esophageal temperature probe will be removed, and the patient extubated after emergence from anesthesia. This will conclude the study and subsequent management will be at the discretion of the attending anesthesiologist

ELIGIBILITY:
Inclusion Criteria:

* Body-mass index 20-36 kg/m2;
* Age 18-75 yrs;
* ASA Physical Status 1-3.

Exclusion Criteria:

* Patient requires an intravenous or arterial catheter distal to the elbow on both arms;
* Serious skin lesions on the hands or arms;
* History of serious vascular disease in the arms;
* Pre-operative fever;
* Contraindication to sevoflurane endotracheal anesthesia.
* Pre-existing neuropathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Warm-water Sleeve: The vital HEAT (vH2) Temperature Management System will be placed on the subject's arm prior to surgery,become activated after anesthesia administration and remain active until surgery ends.
  vital HEAT (vH2) Temperature Management System: The vital HEAT (vH2) Temperature Management System will be placed on the subjects arm prior to surgery. remain on the arm during surgery and removed after surgery.
- Forced Air: Subjects assigned the forced-air warming cover will be positioned over the upper body and exposed arms before surgery begins. The forced-air warmer will be removed when surgery is completed.
  a forced-air warming cover: A forced-air warming cover will be placed on the subject prior to surgery, remain on the subject during surgery and removed after surgery.
Period: Overall Study
Arm/Group | Warm-water Sleeve | Forced Air
Started | 38 | 35
Completed | 37 | 34
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: 5 patients with missing data, including 3 in the warm-water sleeve group and 2 in the forced air group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Warm-water Sleeve | Forced Air | Total
Number analyzed (Participants) | 37 | 34 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (15) | 50 (15) | 49 (15)
Sex/Gender, Customized [Number; unit: participants]
  Female | 11 | 14 | 25
  Male | 23 | 18 | 41
  Missing | 3 | 2 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  White | 32 | 31 | 63
  African American | 1 | 1 | 2
  Unknown | 4 | 2 | 6
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 26.1 (6.6) | 26.3 (5.3) | 26.2 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Distal Esophageal (Core) Temperature
Time Frame: at 1 hour
Measure: Mean (Standard Error); unit: °C
Arm/Group | Warm-water Sleeve | Forced Air
Number analyzed (Participants) | 37 | 34
°C | 35.96 (0.081) | 35.87 (0.085)
Statistical Analysis 1: Comparison: Warm-water Sleeve vs Forced Air; Test type: Non-Inferiority or Equivalence — Non-inferiority delta of 0.5°C; p < 0.0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.091, 95% CI 2-sided [-0.139 to 0.321]

ADVERSE EVENTS:
Arm/Group | Warm-water Sleeve | Forced Air
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/34
Other Adverse Events (participants affected / at risk) | 0/37 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes